CLINICAL TRIAL: NCT01648244
Title: The Use of a Computer Assisted Diabetes Decision Support (CADS) System to Improve Outcomes in Patients With Type 2 Diabetes Who Are Treated by Primary Care Providers
Brief Title: The Use of a Computer Program to Help Primary Care Providers Treat Patients With Type 2 Diabetes
Acronym: CADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alicia L. Warnock, Director, Diabetes Institute, Walter Reed National Military Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 353757
Record Dates: First submitted 2012-07-17; First posted 2012-07-24 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Type II Diabetes Mellitus
Keywords: DM, T2DM, Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Computer-Assisted Decision Support (Experimental): These providers will use the CADS program to treat their enrolled patients.
  Interventions: Other: Computer-Assisted Decision Support

INTERVENTIONS:
Other: Computer-Assisted Decision Support — The CADS software makes a recommendation about what medication changes are appropriate with potential alternates. CADS providers will either "accept" or "reject" the recommendation by the software.Providers with their patients are block randomized into CADS or "Usual Care" for 1 year. Patients associated with a CADS provider will upload their blood glucose data weekly and perform a 7-point glucose profile once per month. They will report major hypoglycemic events and hospitalizations at the time of their quarterly visit. Those getting "usual care" will be seen quarterly and will do self-monitoring of blood glucose and have A1c tests as determined by the provider but no less than twice a year.

SUMMARY:
The primary purpose of this study is to determine whether the use of CADS by primary care providers (PCPs) for their patients with type 2 diabetes (T2DM) changes the quality of care relative to a "usual care" group in terms of objective outcome measures of glycemic control (e.g., A1c, mean blood glucose, frequency of hypoglycemic episodes) and in terms of subjective ratings by patients.

DETAILED DESCRIPTION:
The CADS software integrates the patient's home blood glucose data with appropriate laboratory data (e.g. A1c, liver function, kidney function), demographic data (age, gender), current and previous medications, and active/inactive medical diagnoses. The software makes a recommendation about what medication changes are appropriate with potential alternates. Providers with their patients are block randomized into CADS or "Usual Care" for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Non-specialist physician (general internist or family practitioner), nurse practitioner, physicians assistant
* Absence of orders for deployment or permanent change of station
* Willingness to recruit up to 19 patients prior to randomization
* Willingness to deliver "usual care" as defined in Section 6.3.2 of the protocol.

Exclusion Criteria:

* Specialist physicians
* Orders for deployment or permanent change of station
* Unwillingness to recruit up to 19 patients prior to randomization
* No prior experience with management of type 2 diabetes in adults
* Unwillingness to deliver "usual care" as defined in Section 6.3.2 of the protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in A1c | baseline, 12, 24, 36, and 48 months
  Change is A1c will be measured 5 times over the course of the study to compare the patients for whom the provider is using CADS to those patients whose providers are delivering "usual care".

SECONDARY OUTCOMES:
Major events | ongoing
  The number of major ("severe") hypoglycemic events whether subjective (undocumented) or objective (SMBG or other confirmation, need for intervention, seizure, coma), and emergency room visits for DM-related causes.
Other DM-related events | ongoing
  Number of ER visits for DM-related causes, DM-related hospitalizations and hospital days, and DM-related clinic visits.
Glucose measures | baseline, 12, 24, 36, 48 months
  Mean pre-prandial glucose, mean post-prandial glucose, post-prandial glucose excursions
Blood pressure | baseline, 12, 24, 36, and 48 months
  Clinically significant or statistically detectable changes in BP
Lipids | baseline, 12, 24, 36, and 48 months
  Clinically significant or statistically detectable changes in lipid profile.
Patient satisfaction with treatment | basline and 48 months
  Clinically significant or statistically detectable changes in satisfaction with treatment as measured by the DTSQ.
Quality of life | baseline and 48 months
  Clinically significant or statistically detectable changes in quality of life for patients with DM as measured by the SF-8.
Degree of Acceptance | baseline and 48 months
  The degree of acceptance of CADS by PCPs as measured by a technical assessment questionnaire.
Acceptance of uploading data | baseline, 12, 24, 36, and 48 months
  The degree of acceptance of uploading the glucose meters by patients as measured by a technical assessment questionnaire.
Demographic variables | baseline and 48 months
  The relationship of the primary and/or secondary outcomes to the type of provider, board-certification or eligibility, years in practice, age and gender.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Vigersky, M.D., Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States